CLINICAL TRIAL: NCT01465048
Title: A Pilot Study to Optimise Controlled Human Malaria Infections Using Plasmodium Falciparum Sporozoites Administered by Needle and Syringe
Brief Title: Optimisation of Controlled Human Malaria Infection Using Sporozoites Administered by Needle and Syringe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Sanaria Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: VAC049
Record Dates: First submitted 2011-10-27; First posted 2011-11-04 (Estimated); Results first posted 2013-05-28 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Malaria; Plasmodium Falciparum
Keywords: Malaria; Protozoan Infections; Parasitic Diseases; Malaria Challenge
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Protozoan Infections; Parasitic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plasmodium falciparum sporozoites 2sites (Experimental): 2,500 sporozoites intradermally
  Interventions: Biological: Plasmodium falciparum sporozoites 2sites
- Plasmodium falciparum sporozoites 1 site (Experimental): 2,500 sporozoites intramuscularly
  Interventions: Biological: Plasmodium falciparum sporozoites 1 site
- Plasmodium falciparum sporozoites 1site (Experimental): 25,000 sporozoites intramuscularly
  Interventions: Biological: Plasmodium falciparum sporozoites 1site

INTERVENTIONS:
Biological: Plasmodium falciparum sporozoites 2sites — Aseptic, purified, cryopreserved Plasmodium falciparum sporozoites, 2,500 sporozoites, 50ulx2, 2 intradermal injection sites
  Arms: Plasmodium falciparum sporozoites 2sites
Biological: Plasmodium falciparum sporozoites 1 site — Aseptic, purified, cryopreserved Plasmodium falciparum sporozoites, 2,500 sporozoites, 50ulx2, 2 intramuscular injection sites
  Arms: Plasmodium falciparum sporozoites 1 site
Biological: Plasmodium falciparum sporozoites 1site — Aseptic, purified, cryopreserved Plasmodium falciparum sporozoites, 25,000 sporozoites, 50ulx2, 2 intramuscular injection sites
  Arms: Plasmodium falciparum sporozoites 1site

SUMMARY:
This is an open label, human pilot study to optimise controlled human malaria infection (CHMI) administered by Plasmodium falciparum sporozoites (PfSPZ. Volunteers will be inoculated with PfSPZ Challenge. The route of administration and dose will vary in order to identify the optimal regimen that achieves the greatest infection rate in volunteers with Plasmodium falciparum. All volunteers recruited will be healthy adults aged between 18 and 45 years. Safety and infectivity data will be collected for each of the regimens.

DETAILED DESCRIPTION:
Studies involving CHMI are a powerful tool for investigating malaria vaccine and prophylactic drug efficacy.CHMI has now become established as a key tool to assess the efficacy of novel malaria vaccines and drugs. As CHMI trials are carried out in a controlled environment, they allow unprecedented detailed evaluation of parasite growth and immunological responses, providing essential information for vaccine and drug development.

Out of three currently available methods of performing experimental human malaria infections (blood stage infection, mosquito bites and sporozoite infection), experimental injection directly by needle and syringe using aseptic, purified, cryopreserved sporozoites is, in principle, the most accurate and practical way of dosing sporozoites for challenge studies. Recently, Sanaria Inc have been able to overcome the technical issues associated with the production of aseptic, purified, cryopreserved Plasmodium falciparum sporozoites. As a result, an Investigational New Drug application (IND) was submitted to the U.S. Food and Drug Administration in February 2009, and a Phase 1 clinical trial with experimental challenge of volunteers was initiated in April 2009. Another trial sponsored by Sanaria to find the dose of aseptic, purified, cryopreserved sporozoites that should be used for experimental human malaria infections is currently ongoing with collaboration with the Radboud University Nijmegen Medical Center, The Netherlands.

This trial will be the first time aseptic, purified, cryopreserved P. falciparum sporozoites have been administered intramuscularly to humans.

ELIGIBILITY:
Inclusion Criteria:

* Women only: Must practice continuous effective contraception for the duration of the study.
* Agreement to refrain from blood donation during the course of the study and for at least 3 years after the end of their involvement in the study.
* Written informed consent to undergo CHMI.
* Reachable (24/7) by mobile phone during the whole study period.
* Willingness to take a curative anti-malaria regimen.
* For volunteers not living in Oxford: agreement to stay in a hotel room close to the trial centre during a part of the study (At least Day 6.5 post inoculation until 2 days after treatment commenced).
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

* History of clinical P. falciparum malaria.
* Travel to a malaria endemic region during the study period or within the preceding six months with positive P. falciparum serology at screening.
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrolment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
* Receipt of an investigational product in the 30 days preceding enrollment, or planned receipt during the study period.
* Prior receipt of an investigational malaria vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrollment.
* History of sickle cell anemia, sickle cell trait, thalassemia or thalassemia trait.
* Pregnancy, lactation or intention to become pregnant during the study
* A history of allergic disease or reactions likely to be exacerbated by malaria infection.
* Contraindications to the use of all three proposed anti-malarial medications; Malarone, Riamet and Chloroquine.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrollment.
* Seropositive for hepatitis B surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV).
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.39
* Positive family history in 1st and 2nd degree relatives < 50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, DPhil FRCP, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Mukhopadhyay ES, Bellamy DG, Tinto H, Hamaluba M, Truby A, Salman AM, Hill AVS. Naturally acquired immune responses to alpha-gal in malaria endemic settings and pre-clinical efficacy testing with R21/MM. Vaccine. 2025 Dec 5;68:127897. doi: 10.1016/j.vaccine.2025.127897. Epub 2025 Nov 1. PMID 41176969
- [Derived] Longley RJ, Halbroth BR, Salman AM, Ewer KJ, Hodgson SH, Janse CJ, Khan SM, Hill AVS, Spencer AJ. Assessment of the Plasmodium falciparum Preerythrocytic Antigen UIS3 as a Potential Candidate for a Malaria Vaccine. Infect Immun. 2017 Feb 23;85(3):e00641-16. doi: 10.1128/IAI.00641-16. Print 2017 Mar. PMID 28031267
- [Derived] Hodgson SH, Llewellyn D, Silk SE, Milne KH, Elias SC, Miura K, Kamuyu G, Juma EA, Magiri C, Muia A, Jin J, Spencer AJ, Longley RJ, Mercier T, Decosterd L, Long CA, Osier FH, Hoffman SL, Ogutu B, Hill AV, Marsh K, Draper SJ. Changes in Serological Immunology Measures in UK and Kenyan Adults Post-controlled Human Malaria Infection. Front Microbiol. 2016 Oct 13;7:1604. doi: 10.3389/fmicb.2016.01604. eCollection 2016. PMID 27790201
- [Derived] Sheehy SH, Spencer AJ, Douglas AD, Sim BK, Longley RJ, Edwards NJ, Poulton ID, Kimani D, Williams AR, Anagnostou NA, Roberts R, Kerridge S, Voysey M, James ER, Billingsley PF, Gunasekera A, Lawrie AM, Hoffman SL, Hill AV. Optimising Controlled Human Malaria Infection Studies Using Cryopreserved P. falciparum Parasites Administered by Needle and Syringe. PLoS One. 2013 Jun 18;8(6):e65960. doi: 10.1371/journal.pone.0065960. Print 2013. PMID 23823332

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PfSPZ Challenge 2,500 ID | PfSPZ Challenge 2,500 IM | PfSPZ Challenge 25,000 IM
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PfSPZ Challenge 2,500 ID | PfSPZ Challenge 2,500 IM | PfSPZ Challenge 25,000 IM | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 3 | 3 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Infected
Description: To determine the infectivity rates of PfSPZ Challenge administered in various regimens by thick film microscopy and highly sensitive PCR for Plasmodium falciparum DNA.
Time Frame: 21 days post administration of PfSPZ Challenge
Measure: Number; unit: Participants
Arm/Group | PfSPZ Challenge 2,500 ID | PfSPZ Challenge 2,500 IM | PfSPZ Challenge 25,000 IM
Number analyzed (Participants) | 6 | 6 | 6
Participants | 5 | 3 | 6

2. Secondary Outcome: Frequency, Incidence and Nature of Adverse Events and Serious Adverse Events Arising.
Description: To assess the safety of PfSPZ Challenge administered in various regimens by analysing actively and passively collected data from clinical review of volunteers and laboratory measurements, including lab reports and adverse events.
Time Frame: Participants will be followed for the duration of the study, an expected average of 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Dynamics of Plasmodium Falciparum Parasite Growth Following PfSPZ Challenge Administered in Various Regimens
Description: To determine the parasite growth dynamics of PfSPZ Challenge administered in various regimens using highly sensitive PCR for Plasmodium falciparum DNA.
Time Frame: 21 days post administration of PfSPZ Challenge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 07/11/11 to 13/02/12
Arm/Group | PfSPZ Challenge 2,500 ID | PfSPZ Challenge 2,500 IM | PfSPZ Challenge 25,000 IM
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PfSPZ Challenge 2,500 ID (N=6) | PfSPZ Challenge 2,500 IM (N=6) | PfSPZ Challenge 25,000 IM (N=6)
Headache (General disorders) | 2 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Malasie (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gum Bleeding (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No